CLINICAL TRIAL: NCT05937568
Title: Expanded Access Treatment With Imetelstat For Adult Participants With Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS) Who Are Transfusion-Dependent And Have Failed to Respond or Have Lost Response or Are Ineligible For Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: Expanded Access for Treatment With Imetelstat
Status: Approved for marketing | Type: Expanded Access
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MDSEAP001
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — imetelstat

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Imetelstat — Participants will receive imetelstat, intravenously (IV) by infusion every 4 weeks.

SUMMARY:
The objective of this expanded access protocol (EAP) is to provide access to treatment with imetelstat, the Investigational Product (IP), for eligible adult participants diagnosed with very low, low, intermediate risk (by Revised International Prognostic Scoring System, IPSS-R) myelodysplastic syndromes (MDS) who are red blood cell (RBC) transfusion-dependent, have failed to respond or have lost response or are ineligible for ESAs, had not received prior treatment with either a hypomethylating agent or lenalidomide and were non-del(5q), until such time that imetelstat becomes commercially available.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of MDS according to World Health Organization (WHO) criteria confirmed by bone marrow aspirate and/or biopsy preferably within 24 but no more than 52 weeks prior to EAP start.
* Very Low, Low, or Intermediate risk MDS (≤3.5) per IPSS-R.
* Red blood cell (RBC) transfusion dependent, defined as requiring at least 4 RBC units over an 8-week period during the 16 weeks prior to EAP entry; pre-transfusion hemoglobin (Hb) should be less than or equal to 9.0 grams per deciliter (g/dL) to count towards the 4 units total.
* Has MDS that has failed to respond or has lost response or are ineligible for ESAs.
* To ensure participants have adequate iron stores they must have transferrin saturation greater than 20% and serum ferritin greater than 400 nanograms per milliliter (ng/mL).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
* Hematology and biochemical laboratory test values within the protocol defined limits.
* Have no approved alternative treatment available.
* Inability to participate in a current imetelstat clinical study for the disease or conditions.
* Have a treating physician who has appropriately evaluated the benefit/risk profile for potential imetelstat treatment.

Key Exclusion Criteria:

* Have previously assessed as having IPSS-R high or very high risk MDS.
* Participant with del(5q) karyotype.
* Participant with MDS/myeloproliferative neoplasm Overlap Syndromes.
* Participant has known allergies, hypersensitivity, or intolerance to imetelstat or its excipients.
* Participant has received an experimental or investigational product or used an invasive investigational medical device within 30 days prior to EAP entry or is currently enrolled in an investigational study.
* Prior treatment with imetelstat; or eligible for enrollment in an ongoing imetelstat clinical trial.
* Prior treatment with lenalidomide or a hypomethylating agent (example, azacitidine, decitabine, or decitabine/cedazuridine).
* Has received an ESA or any anti-MDS therapy, chemotherapy, immunomodulatory, or immunosuppressive therapy within 4 weeks prior to EAP entry.
* Prior history of hematopoietic stem cell transplant.

Note: Other protocol specified inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult